CLINICAL TRIAL: NCT02944357
Title: Pilot Study of Gemcitabine and Cisplatin Plus AGS-003-BLD in Patients With Muscle-Invasive Bladder Cancer Undergoing Neoadjuvant Cisplatin-Based Chemotherapy
Brief Title: Gemcitabine Hydrochloride, Cisplatin, and AGS-003-BLD in Treating Patients With Muscle-Invasive Bladder Cancer Undergoing Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1452; NCI-2016-01517 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1452 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2016-10-19; First posted 2016-10-25 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2016-10

CONDITIONS: Infiltrating Bladder Urothelial Carcinoma; Stage II Bladder Urothelial Carcinoma; Stage III Bladder Urothelial Carcinoma; Stage IV Bladder Urothelial Carcinoma
MeSH Terms: interventions — Cisplatin; transplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gemcitabine; Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (gemcitabine hydrochloride, cisplatin, AGS-003-BLD) (Experimental): NEOADJUVANT PHASE: Patients receive gemcitabine hydrochloride IV on days 1 and 8, AGS-003-BLD ID on day 1, and cisplatin IV on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive AGS-003-BLD ID on day 1. Treatment repeats every 14 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  SURGERY: Patients undergo cystectomy during course 8.
  ADJUVANT PHASE: Patients continue AGS-003-BLD ID on day 1 of course 9. Treatment repeats every 12 weeks for up to 9 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine Hydrochloride; Procedure: Radical Cystectomy; Biological: Tumor Cell-Derived Vaccine Therapy

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroamine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP (diamminedichloroplatinum); Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011; LY188011
Procedure: Radical Cystectomy — Undergo cystectomy
  Other Names: Complete Cystectomy
Biological: Tumor Cell-Derived Vaccine Therapy — Given AGS-003-BLD ID

SUMMARY:
This pilot clinical trial studies how well gemcitabine hydrochloride, cisplatin, and AGS-003-BLD work in treating patients with bladder cancer that has spread to the muscle and who are undergoing surgery. Drugs used in chemotherapy, such as gemcitabine hydrochloride and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Vaccines made from a person's tumor cells may help the body build an effective immune response to kill tumor cells. Giving gemcitabine hydrochloride, cisplatin, and AGS-003-BLD before surgery may make the tumor smaller and reduce the amount of tissue that needs to be removed by surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the immunogenicity of AGS-003-BLD in subjects with muscle invasive bladder cancer.

SECONDARY OBJECTIVES:

I. To assess 1-year disease-free survival rate of patients with muscle-invasive bladder cancer who receive cisplatin/gemcitabine chemotherapy plus AGS-003-BLD.

II. To determine the time to first metastatic lesion. III. To explore the disease-free and overall survival of patients treated with this treatment combination.

IV. To evaluate the pathologic complete response (pCR) rate and identify any activity of this treatment combination.

V. To evaluate toxicities and tolerability associated with this treatment combination.

VI. To assess the success rate of tumor procurement and AGS-003-BLD production of >= 5 doses.

TERTIARY OBJECTIVES:

I. To evaluate the relationships between pathologic complete response with the change in CD28+ T cell levels.

II. To evaluate the change in frequency of CD11a highPD-1+ CD8+ T cells (and their expression of Bim) in peripheral blood.

OUTLINE:

NEOADJUVANT PHASE: Patients receive gemcitabine hydrochloride intravenously (IV) on days 1 and 8, AGS-003-BLD intradermally (ID) on day 1, and cisplatin IV on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive AGS-003-BLD ID on day 1. Treatment repeats every 14 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

SURGERY: Patients undergo cystectomy during course 8.

ADJUVANT PHASE: Patients continue AGS-003-BLD ID on day 1 of course 9. Treatment repeats every 12 weeks for up to 9 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION INCLUSION CRITERIA: Diagnosis or clinical signs of urothelial carcinoma with clinical stage T2 or greater disease without lymph node involvement where neoadjuvant chemotherapy of cisplatin and gemcitabine are indicated
* PRE-REGISTRATION INCLUSION CRITERIA: Scheduled for a transurethral resection of bladder tumor (TURBT)
* PRE-REGISTRATION INCLUSION CRITERIA: Be a candidate for radical cystectomy
* PRE-REGISTRATION INCLUSION CRITERIA: Signed and dated informed consent document for study participation
* PRE-REGISTRATION INCLUSION CRITERIA: Willing to submit tissue for required correlative research
* REGISTRATION INCLUSION CRITERIA
* TURBT successfully completed
* Verification received from Argos Therapeutics that ribonucleic acid (RNA) successfully collected from TURBT procedure
* Be a candidate for radical cystectomy
* Diagnosis of urothelial carcinoma with stage T2 or greater disease without lymph node involvement where neoadjuvant chemotherapy of cisplatin and gemcitabine are indicated
* Absolute neutrophil count (ANC) >= 1500/uL
* Platelet count >= 100,000/uL
* Total bilirubin =< 1.5 x institutional upper normal limit (UNL) or =< 3 x institutional UNL if known Gilbert's syndrome
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x UNL
* Alkaline phosphatase =< 5 x UNL
* Hemoglobin >= 9.0 g/dL
* International normalized ratio (INR) and partial thromboplastin time (PTT) =< 3.0 x UNL; NOTE: anticoagulation is allowed if target INR =< 3.0 x UNL on a stable dose of warfarin or on a stable dose of low molecular weight heparin for > 2 weeks at time of registration
* Calculated creatinine clearance must be >= 50 ml/min using the applicable Cockcroft-Gault formula
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Ability to provide written informed consent
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Willing to provide tissue and blood samples for correlative research purposes
* Negative serum pregnancy test for female subjects with reproductive potential =< 7 days prior to registration, for women of childbearing potential only
* Able to abstain from taking prohibited drugs, either prescription or non-prescription, during the treatment phase of the study

Exclusion Criteria:

* RE-REGISTRATION EXCLUSION CRITERIA
* Requirement for systemic chronic immunosuppressive drugs or systemic chronic corticosteroids for active autoimmune disorder(s) or other conditions (e.g.: rheumatoid arthritis, systemic lupus erythematous, multiple sclerosis, organ transplant recipient, etc.)
* Known inability to undergo neoadjuvant gemcitabine and cisplatin combination treatment due to pre-existing medical conditions in the opinion of the treating physician or investigator
* Immunotherapy =< 28 days prior to pre-registration (e.g. intravesical Bacillus Calmette-Guerin [BCG])
* Any of the following prior therapies:

  * Systemic chemotherapy for bladder cancer at any time; NOTE: intravesical chemotherapy is allowed
  * Systemic chemotherapy for other malignancies =< 3 years prior to pre-registration
* REGISTRATION EXCLUSION CRITERIA
* Lymph node positive urothelial carcinoma
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements in the opinion of the investigator
* Treatment with oral/systemic corticosteroids =< 14 days prior to registration, with the exception of topical or inhaled steroids or steroids given for the purpose of antiemetics during chemotherapy
* New York Heart Association classification III or IV congestive heart failure
* Central nervous system (CNS) metastases or seizure disorder
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation) with the exception of intravesical therapy at the time of TURBT
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Clinically significant infections including human immunodeficiency virus (HIV), syphilis, and active hepatitis B or C
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Prior history of malignancy =< 3 years prior to registration, except for adequately treated non-melanoma skin cancer, adequately treated early stage breast cancer, adequately treated cervical cancer and non-metastatic prostate cancer under clinical control as deemed by treating physician or investigator
* History of myocardial infarction =< 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* History of major surgery or traumatic injury =< 28 days prior to registration or other major anticipated procedures requiring general anesthesia during study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2017-09-05 (Actual)

PRIMARY OUTCOMES:
Change in the frequency of CD11a high PD-1+ CD8+ T cells | Baseline, before systemic therapy with chemotherapy
  Descriptive statistics (mean, standard deviation [sd], median, interquartile range [iqr]) will be used to summarize change from baseline in the frequency of CD11a high PD-1+ CD8+ T cells following five doses of AGS-003-BLD.
Change in the frequency of CD11a high PD-1+ CD8+ T cells | Prior to 1st dose of AGS-003-Bladder therapy
  Descriptive statistics (mean, standard deviation [sd], median, interquartile range [iqr]) will be used to summarize change from baseline in the frequency of CD11a high PD-1+ CD8+ T cells following five doses of AGS-003-BLD.
Change in the frequency of CD11a high PD-1+ CD8+ T cells | Treatment visit 7 (Cycle 3) After 3rd dose of AGS-003-Bladder therapy, up to 7 days
  Descriptive statistics (mean, standard deviation [sd], median, interquartile range [iqr]) will be used to summarize change from baseline in the frequency of CD11a high PD-1+ CD8+ T cells following five doses of AGS-003-BLD.
Change in the frequency of CD11a high PD-1+ CD8+ T cells | Treatment visit 15 (Cycle 6) - After the 5th dose of neoadjuvant AGS-003-Bladder therapy, up to 14 days
  Descriptive statistics (mean, standard deviation [sd], median, interquartile range [iqr]) will be used to summarize change from baseline in the frequency of CD11a high PD-1+ CD8+ T cells following five doses of AGS-003-BLD.
Change in the frequency of CD11a high PD-1+ CD8+ T cells | Treatment visit 20 (Cycle 8) - After the 8th dose (3rd adjuvant) of AGS-003 - Bladder therapy, up to 12 weeks
  Descriptive statistics (mean, standard deviation [sd], median, interquartile range [iqr]) will be used to summarize change from baseline in the frequency of CD11a high PD-1+ CD8+ T cells following five doses of AGS-003-BLD.

SECONDARY OUTCOMES:
1-year survival rate | 1 year
2-year disease-free survival rate | 2 years
2-year survival rate | 2 years
Disease-free survival rate | 1 year
Incidence of adverse events assessed by National Cancer Institute Common Terminology Criteria for Adverse Events | Up to 2 years
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine adverse event patterns.
Manufacturing success rate and successful manufacture of > 5 doses and administration of 1 or more doses of AGS-003-BLD | Up 2 years
  Descriptive statistics (frequency table) and histogram will be used to summarize the success rate.
Proportion of pathologic complete responses | Up to 2 years
  Descriptive statistics (frequency table) and histogram will be used to summarize the pathologic complete response rate.
Time to first metastatic lesion | Time from randomization to first recognition of metastases, assessed up to 2 years
  Will be estimated using the Kaplan-Meier method.

OTHER OUTCOMES:
Change in CD28 + T cell level with pathological complete response | Baseline up to 2 years
  Descriptive statistics (mean, sd, median, iqr) and longitudinal plots (raw value, change, and change in percentage) will be used to summarize the correlative endpoints. Further analysis will depend on the amount of data received and will be mainly exploratory.
Change in frequency of CD11a high PD-1+ CD8+ T cells (and their expression of Bim) in peripheral blood | Baseline up to 2 years
  Descriptive statistics (mean, sd, median, iqr) and longitudinal plots (raw value, change, and change in percentage) will be used to summarize the correlative endpoints. Further analysis will depend on the amount of data received and will be mainly exploratory.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Costello, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States